CLINICAL TRIAL: NCT04075565
Title: The Psychophysiological Effect of Simulated and Terrestrial Altitude
Acronym: Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Collaborators: University of Portsmouth (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-00504
Record Dates: First submitted 2019-08-07; First posted 2019-08-30 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Hypoxia; Altitude Hypoxia; Altitude Sickness; Altitude; Mountain Sickness; Hypoxia, Altitude
Keywords: hypoxia; altitude; physiology; cognition
MeSH Terms: conditions — Hypoxia; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: The study design is a crossover design.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simulated altitude (Active Comparator): The participants are exposed to simulated altitude in a normobaric situation.
  Interventions: Behavioral: Cloud 9
- Terrestrial altitude (Experimental): The participants are exposed to terrestrial altitude in a hypobaric situation.
  Interventions: Behavioral: Terrestrial altitude
- Control (No Intervention): the participants are exposed to a normoxic and normobaric environment.

INTERVENTIONS:
Behavioral: Terrestrial altitude — Terrestrial altitude: The volunteers are in an SAC hut at an altitude of 3000 m. By means of this exposure the psychophysiological effect under hypobaric and hypoxic conditions is determined. The subjects spend the night in this SAC hut and the measurements are repeated the next day.
  Arms: Terrestrial altitude
Behavioral: Cloud 9 — Cloud 9 is a solid, certified product that complies with European Directives on Electromagnetic Compatibility, Machine Directive, Air Pressure Equipment and Low Voltage Equipment (89/336 / EEC, 91/368 / CEE, 93/68 / CEE, 97/23 / EC, EN61010-1 All directives are in writing in the Supplements to this Ethics Application.
  Simulated height: The subjects are in the laboratory of our institution and are connected to the Cloud 9 by means of a mask. Subjects are exposed to a simulated altitude of 3530m under normobaric conditions. By means of this intervention the psychophysiological effect under normobaric and hypoxic conditions is determined.
  Arms: Simulated altitude

SUMMARY:
The aim of this study is to compare the psychophysiological effects of terrestrial altitude with a normobaric, hypoxic situation.

DETAILED DESCRIPTION:
Research has consistently shown that exposure to extreme environments (such as high altitude stays) may affect cognitive function. For logistical reasons and to control the experimental set-ups, most of these examinations are carried out in the laboratory. By testing under such controlled conditions, researchers can remove any co-foundational factors and isolate the cause of stress, thereby better understanding the mechanisms by which impairment can occur. However, when people are exposed to such environments in the "real world" (such as altitude), they often experience a number of other additional stressors at the same time, which can also affect their performance. Surprisingly, however, little attention has been paid to the study of these additional stressors in combination.

Although the oxygen content remains constant at various altitudes (20.93%), the air pressure decreases exponentially as the altitude increases. As a result, the oxygen partial pressure in arterial blood and tissue is reduced (hypoxia), leading to a deterioration in both physical and cognitive performance. Hypoxic conditions also alter the perception of pain, which may be particularly relevant for patients suffering from hypoxic conditions. According to the authors' knowledge, there is limited literature investigating and comparing simulated and real psychophysiological responses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adults aged 18 to 50 years
* No cardiovascular disease and / or surgery
* no surgery on the cardiovascular system.
* No current injuries and / or pain
* Regular and adequate sleep
* No terrestrial altitude of 1000 m exceeded last month (including flights)
* No form of hypoxia exposed last month

Exclusion Criteria:

* Age over 50 years
* current injuries of any kind and / or pain
* Acute and / or chronic pain conditions Known general diseases (e.g., diabetes mellitus)
* fear of hypoxia
* fear of heights or sensitivity to terrestrial altitude
* Regular use of medicines (also bought by yourself), except for contraceptives
* Cardiovascular diseases or abnormalities
* Anomalies of the blood analysis or ECG
* Psychological disorders
* pregnancy / lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Perfusion of the skin microcirculation | 30 minutes
  Perfusion of skin microcirculation is demonstrated non-invasively using the Laser Speckle Contrast Imager (moorFLPI 2, moor instruments, www.moor.co.uk). This measurement is taken during the baseline measurements, after the step-up task and up to 30 minutes after the cold water bath of the hand (5 minute interval). This outcome measure reports the change from baseline for the perfusion of the skins' microcirculation.
Oxygenation of the muscles and the brain | 30 minutes
  Muscle and brain oxygen saturation is measured non-invasively using a deep tissue oxygenation monitor (moorVMS-NIRS, moor instruments, www.moor.co.uk). For this purpose, adhesive electrodes are applied over the muscle and the forehead. This measurement is taken during the baseline measurements, after the step-up task and up to 30 minutes after the cold water bath of the hand (5 minute interval). This outcome measure reports the change from baseline for the oxygenation of the muscles and the brain.
Oxygenation of the blood | 30 minutes
  The oxygen saturation of the blood is measured with a portable pulse oximeter with finger clip probe (Nonin 7500, Nonin medical B.V., Plymouth, USA). This measurement is taken during the baseline measurements, after the step-up task and up to 30 minutes after the cold water bath of the hand (5 minute interval). This outcome measure reports the change from baseline for the oxygenation of the blood.
Blood pressure | 30 minutes
  Blood pressure (systolic and diastolic) is detected by an electronically automated upper arm blood pressure monitor (Boso-Medicus uno). This measurement is taken during the baseline measurements, after the step-up task and up to 30 minutes after the cold water bath of the hand (5 minute interval). This outcome measure reports the change from baseline for the blood pressure.
Heart rate | 30 minutes
  The heart rate is measured using a pulse belt and an additional 2-point ECG (Actiheart, Camntech Ltd., Cambridge, UK). This measurement is taken during the baseline measurements, after the step-up task and up to 30 minutes after the cold water bath of the hand (5 minute interval). This outcome measure reports the change from baseline for the heart rate.
Skin temperature | 30 minutes
  Skin temperature is measured using the iButton system (www.ibuttonlink.com). The self-adhesive sensors wirelessly transmit skin temperature information to a computer. Furthermore, the skin temperature is recorded by means of a thermal imaging camera (FLIR). This measurement is taken during the baseline measurements, after the step-up task and up to 30 minutes after the cold water bath of the hand (5 minute interval). This outcome measure reports the change from baseline for the skin temperature.
Concentration of blood lactate and creatine kinase | 30 minutes
  Lactate and creatine kinase measurements are performed by capillary blood measurement (Accutrend, Roche Diagnostic, Red Cross, Switzerland & Reflotron, Roche Diagnostic, Rotkreuz, Switzerland). This measurement is taken during the baseline measurements, after the step-up task and up to 30 minutes after the cold water bath of the hand (5 minute interval). This outcome measure reports the change from baseline for lactate and creatine kinase.
Balance | 30 minutes
  The fluctuations of the hull are recorded and evaluated with the Sway Star Systems (www.b2i.info). The Sway Star is a measuring instrument that contains gyroscopes. It is attached to a strap which is applied around the waist of the patient. The data is evaluated with the associated Sway Star software and transferred to the data sheet. This measurement is performed after the baseline measurement and after the cold water bath immersion of the hand. This outcome measure reports the change from baseline for balance.
Pain threshold: pain pressure gauge | 30 minutes
  The pain threshold is measured by means of a pain pressure gauge (NOD, www.to-nod.com). This measurement is performed after the baseline measurement and after the cold water bath immersion of the hand. This outcome measure reports the change from baseline for pain threshold.
Sleep disorder | 30 minutes
  Sleep disorder is measured with "Standford sleepiness scale", choosing one answer from seven (1=no sleepiness, 7=extreme sleepiness). The measurements are performed at baseline and after the cold water bath immersion of the hand and report the change from baseline.
Altitude sickness | 30 minutes
  Altitude sickness is measured with "Lake Louis acute mountain sickness scale", choosing the most appropriate answer from 5 questions. Questions range from 0 (=no symptoms) to 4 (=severe symptoms).The measurements are performed at baseline and after the cold water bath immersion of the hand and report the change from baseline.
Dyspnoea | 30 minutes
  Dyspnoea is measured with the "modified BORG scale", choosing a number from 0 (=no dyspnoea) to 10 (=maximum dyspnoea). The measurements are performed at baseline and after the cold water bath immersion of the hand and report the change from baseline.
Mental state | 30 minutes
  Mental state is assessed using "profile of the mood state", answering 37questions. Each question has a score from 0 (=not at all) to 4 (=extremely). The total sum of the scores is used. The measurements are performed at baseline and after the cold water bath immersion of the hand and report the change from baseline.
Cognition | 30 minutes
  Cognitive tests consists of 8 tasks (automated neuropsychological assessment metrics). Lower values are better than higher values and are analyzed individually. The measurements are performed at baseline and after the cold water bath immersion of the hand and report the change from baseline.

SECONDARY OUTCOMES:
Thermal comfort and sensation | 30 minutes
  These parameters are measured by a thermal comfort scale (ranging from 0 [comfortable] to +4 [very uncomfortable]) and a thermal sensation scale (ranging from -4 [ver cold] to +4 [very hot]). These measurements are performed after the baseline measurement and after the cold water bath immersion of the hand and report the change from baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Fachhochschule Südschweiz, Landquart, Kanton Graubünden
  - Fachhochschule Südschweiz, Landquart

IPD SHARING:
Plan to Share IPD: No